CLINICAL TRIAL: NCT01584323
Title: Pomegranate to Reduce Maternal and Fetal Oxidative Stress and Improve Outcome in Pregnancies Complicated With Preterm Premature Rupture of the Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yuval Ginsberg, MD, M.D, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0231-11-RMB
Record Dates: First submitted 2012-04-16; First posted 2012-04-24 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Preterm Premature Rupture of Membranes; Pregnant State
Keywords: Preterm premature rupture of membranes; pomgranate; oxidative stress; pregnant women with Preterm premature rupture of membranes
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pomegranate pills (Active Comparator): treatment with pomgranate pills to women suffering preterm premature rupture of membranes
  Interventions: Dietary Supplement: Pomgranate pills
- placebo pills (Placebo Comparator): treatment with placebo to women with preterm premature rupture of membranes
  Interventions: Dietary Supplement: Placebo pills

INTERVENTIONS:
Dietary Supplement: Pomgranate pills — Treatment arm will receive The POMx pomegranate 1,000 mg capsule a day for maximum of two weeks or until they deliver if occurs before
  The POMx pomegranate 1,000 mg capsule contains at least 800 mg natural polyphenol using a pomegranate polyphenol standard and is comparable to mg/8 oz juice.(attached is confirmation Similarity of Pomegranate Juice and POMx Polyphenols)
  Arms: Pomegranate pills
Dietary Supplement: Placebo pills — The placebo group will receive placebo pills , for maximum of two weeks or until they deliver if occurs before The palecbo capsule contains gelatin and lactose. The capsuls are manufactured by the hospital pharmacy.All the components are medically approved fot use during pregnancy
  Arms: placebo pills

SUMMARY:
In this study the investigators sought to determine the effects of Pomegranate (Natural pomegranate polyphenol (P. granatum L) extract) :

1. On the maternal and fetal oxidative stress and inflammation associated with PPROM.
2. On the time interval from PPROM to delivery and on fetal Ph and apger score.

DETAILED DESCRIPTION:
Preterm premature rupture of membranes is the rupture of membranes during pregnancy before 37 weeks' gestation. It occurs in 3 percent of pregnancies and is the cause of approximately one third of preterm deliveries. It can lead to significant perinatal morbidity, including respiratory distress syndrome, neonatal sepsis, umbilical cord prolapse, placental abruption, and fetal death.(ref) It increases the risk of prematurity and leads to a number of other perinatal and neonatal complications, including a 1 to 2 percent risk of fetal death.(2) The latent period, which is the time from membrane rupture until delivery, generally is inversely proportional to the gestational age at which PROM occurs. For example, one large study (3) of patients at term revealed that 95 percent of patients delivered within approximately one day of PROM, whereas an analysis of studies(4) evaluating patients with preterm PROM between 16 and 26 weeks' gestation determined that 57 percent of patients delivered within one week, and 22 percent had a latent period of four weeks Numerous risk factors are associated with preterm premature rupture of membrane, lower socioeconomic status, are smokers, have a history of sexually transmitted infections, have had a previous preterm delivery, have vaginal bleeding, or have uterine distension (e.g., polyhydramnios, choriodecidual infection, in many cases the PPROM is associated inflammatory process and increased oxidative stress. Intrauterine inflammation may be associated with, fetal injury preterm birth, low birth weight, and cerebral palsy (5,6,7,8,9). While treatment for PPROM Includes antibiotics it does not aimed to cope with the increased oxidative stress and inflammation that are associated with PPROM and are thought to play important role in the fetal injury Pomegranate juice contains a high concentration of vitamins (C, B1, B2, B3, B5), potassium, Magnesium, Zinc and is a good source for polyphenols (10). Polyphenols molecules have been found to possess antioxidant properties as well as effects on gene expression (11). Recent studies indicate that among foods that contain polyphenols, juice extracted from the pomegranate has the highest concentration of measurable polyphenols (12,13). Pomegranates have shown activity against the cytokine NF-κB and the MAP kinases JNK and ERK, which are critical steps in the cascade of events leading to inflammatory response The NF- κB pathway is activated in response to bacterial infection, and this may explain the effects against bacterial infection (14). Juice consumption may also inhibit viral infection (15).

In a rat animal model pomegranate juice that was given to the dams during pregnancy and lactation period was found as neuroprotective agent to the neonatal mouse brain.(16). Recently Tuuli et al published abstract at the annual meeting of the society of maternal fetal medicine 2011, demonstrating that pomefranate juice (8 oz a day) supplement for the last two weeks to pregnancy, reduced significantly the placental oxidative stress associated with delivery compared to control.

Enhancing the activity or the availability of antioxidants may modulate the inflammatory response associated with PPROM, thereby reducing oxidative stress and the risk to the fetus. In this study we sought to determine the effects of Pomegranate 1. on the maternal and fetal oxidative stress and inflammation associated with PPROM 2. On the time interval from PPROM to delivery and on fetal Ph and apger score.

Study protocol:

All the women admitted with PPROM will receive the usual protocol of the department (Penibrin for two days and Erythromycin for five days)

After signing approval to participate in the study, blood will be drawn for determining the oxidative stress markers (will be analyzed after delivery). The patient will continue the department routine PPROM protocol.

After admission the women will be divided to two groups. One group will receive The POMx pomegranate 1,000 mg capsule a day. The other group will receive placebo. Both groups will receive regiments for a maximum of two weeks or until they deliver if occurs beforehand.

The POMx pomegranate 1,000 mg capsule contains at least 800 mg natural polyphenol using a pomegranate polyphenol standard and is comparable to mg/8 oz juice.(attached is confirmation Similarity of Pomegranate Juice and POMx Polyphenols)

The palecbo capsule contains gelatin and lactose. The capsuls are manufactured by the hospital pharmacy.All the components are medically approved fot use during pregnancy.

During pregnancy:

The patient will continue their usual PPROM protocol.

After delivery After delivery of the baby 1.umbilical blood will be drawn from the umbilical cord and maternal serum for oxidative stress markers Ph and C-reactive protein 2. Histological evaluation of the placenta for inflammation

ELIGIBILITY:
Inclusion Criteria:

* pregnancy
* singleton pregnancy
* preterm premature rupture of membranes
* gestational age > 24Wks

Exclusion Criteria:

* gestational age > 24wks
* fetal anomalies

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Oxidative Stress | Measurments will be first taken at the day of admission (for the mother) and will be assessed immediatly after delivery (mother and newborn)
  Serum lipid peroxidation
  1. Serum lipids peroxidation
  2. Lipid peroxide formation
  3. Paraoxonase activity measurements

SECONDARY OUTCOMES:
Obstetrical outcomes | Measurments will be first taken at the day of admission (for the mother) and will be assessed immediatly after delivery (mother and newborn)
  1. Apgar score
  2. cord PH
  3. cord CRP levels

CONTACTS AND LOCATIONS:
Overall Officials: Ido Solt, M.D, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel